CLINICAL TRIAL: NCT02353767
Title: Evaluation of Liver Fibrosis in HIV-infected Patients With Metabolic Syndrome
Acronym: METAFIB
Status: Completed | Type: Observational
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Sponsor
Other Study IDs: IMEA 42
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Abdominal Obesity Metabolic Syndrome; HIV; Liver Fibrosis
MeSH Terms: conditions — Abdominal obesity metabolic syndrome; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Presence of metabolic syndrome according to the International Diabetes Foundation (IDF)
  Interventions: Procedure: Noninvasive evaluation of liver fibrosis and steatosis
- Controls: * age ± 7 years from cases
  * duration of HIV-1 infection ± 3 years from cases
  * HIV-1 viral load matched to cases according to 3 thresholds: 50 - 500, 501 - 1000 or > 1000 copies/mL
  Interventions: Procedure: Noninvasive evaluation of liver fibrosis and steatosis

INTERVENTIONS:
Procedure: Noninvasive evaluation of liver fibrosis and steatosis — Transient elastography (using the Fibroscan, CAP Fibroscan) and biomarker panels (FibroTest, Fibromètre, Hepascore, Steatotest, Nashtest)

SUMMARY:
This study aims to estimate the prevalence of bridging liver fibrosis and cirrhosis (METAVIR score ≥ F2) according to METAVIR score in HIV infected patients not chronically infected by viral hepatitis but exhibiting a metabolic syndrome according to the IDF definition (International Diabetes Foundation).

DETAILED DESCRIPTION:
HIV-associated morbidity and mortality has been considerably modified ever since the availability of potent antiretroviral treatment in 1996. Recent studies have shown the impact of treatment, with the decreased frequency of AIDS-related diseases coinciding with the preponderance of non-AIDS related pathologies.

Consequently, diseases of hepatic origin have become a key problem in the therapeutic course of HIV-infected patients, representing a major source of significant morbidity and mortality. Liver-related diseases comprise of various etiologies, including co-infection with chronic viral hepatitis and excessive alcohol consumption. When excluding these particular diseases, fibrotic patients exhibit an elevated prevalence of metabolic syndrome, regardless of lipodystrophy. Directly linked to metabolic syndrome, non-alcoholic hepatic steatosis has the capacity to induce necro-inflammatory lesions with an increased risk of evolving into cirrhosis and its complications thereto (i.e. hepatocellular carcinoma, liver decompensation, and end-stage liver disease). In the context of HIV, very little data is available concerning the link between metabolic syndrome and hepatic fibrosis, despite the increasing risk of developing such disease during extended life-span, the long-term disruption of glycolipid metabolism induced by antiretroviral treatment, and the presence of various social risk-factors (i.e. increasing trends in weight gain and decreased physical activity).

The principal objective of the present study is to then characterize the prevalence and determinants associated with hepatic fibrosis among HIV-infected patients, without co-infection with other hepatitis viruses, and who present symptoms of metabolic syndrome according to the AHA 2009 definition. In order to more appropriately answer this research question, we will conduct a nested, matched case-control study including 300 HIV-infected patients per group. We will also aim to identify risk-factors of liver fibrosis other than metabolic syndrome, to study agreement in 4 non-invasive scores of liver fibrosis and 3 non-invasive score of steatosis, and to evaluate the performance of the Controlled Attenuation Parameter (CAP) method for use in diagnosing hepatic steatosis.

All patients in this study will be recruited in a clinical center situated in the infectious disease unit at Saint-Antoine Hospital, where 3400 HIV-infected patients have regular consultations. Patients will be identified from an in-house informatics platform, serving as a surveillance tool for metabolic syndrome, among other diseases, with the intention of increasing better-adapted clinical and therapeutic care. Each patient presenting with metabolic syndrome will be matched with a control patient on the following characteristics: age (±5 years), duration of HIV-infection (±2 years), HIV-RNA viral load (in categories of <50-500, 501-1000, or >1000 copies/mL), and gender. Patients with abnormal transaminases will be excluded from this study.

This study will bring about a clearer understanding of the frequency and importance of liver fibrosis risk in patients with metabolic syndrome, which will allow us to determine the more important elements of surveillance necessary in the prevention and development of hepatic lesions. Accordingly, this study will add more pertinent information regarding treatment guidelines specific to this patient population.

ELIGIBILITY:
Inclusion Criteria:

A. For all patients:

* >18 years of age
* HIV-1 infection for a minimum of 5 years confirmed by Western Blot or ELISA
* Signed and full comprehension of informed consent
* Affiliation to Sécurité Sociale

B. Specific to Cases :

Presence of metabolic syndrome according to the International Diabetes Foundation (IDF)

C. Matched Criteria specific to controls :

* Same age ± 7 years
* Same duration of HIV-1 infection ± 3 years
* Same criterion of HIV-1 viral load (according to 3 thresholds: 50 - 500, 501 - 1000 or > 1000 c/mL)

Exclusion Criteria:

* Chronic hepatitis B (HBs-Ag positive or isolated positive antiHBc-Ab with positive HBV-DNA)
* Chronic hepatitis C (positive antiHCV-Ab)
* Active IV or oral drug use and/or ongoing substitution therapy
* Other known chronic hepatitis : auto-immune hepatitis, primary or secondary biliary cirrhosis, hemochromatosis, Wilson disease, alpha 1 anti-trypsin deficit, primary or secondary sclerosing cholangitis, biliary obstruction, liver vascular disease associated with HIV infection, biliary or liver cancer
* CD4 < 50/mm3
* Any current opportunistic infection
* Serious condition influencing vital status
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients followed in the Infectious Diseases department of Saint-Antoine hospital.
Sampling Method: Non-Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Liver fibrosis | One time
  Liver fibrosis as measured by Fibroscanner

SECONDARY OUTCOMES:
Liver steatosis | One time
  Sub group of patients who had IRM measurements
Hand osteoarthritis | One time
  Sub group of patients who had an X-Ray of their hands

REFERENCES:
- [Background] Lewden C, May T, Rosenthal E, Burty C, Bonnet F, Costagliola D, Jougla E, Semaille C, Morlat P, Salmon D, Cacoub P, Chene G; ANRS EN19 Mortalite Study Group and Mortavic1. Changes in causes of death among adults infected by HIV between 2000 and 2005: The "Mortalite 2000 and 2005" surveys (ANRS EN19 and Mortavic). J Acquir Immune Defic Syndr. 2008 Aug 15;48(5):590-8. doi: 10.1097/QAI.0b013e31817efb54. PMID 18645512
- [Background] Worm SW, Friis-Moller N, Bruyand M, D'Arminio Monforte A, Rickenbach M, Reiss P, El-Sadr W, Phillips A, Lundgren J, Sabin C; D:A:D study group. High prevalence of the metabolic syndrome in HIV-infected patients: impact of different definitions of the metabolic syndrome. AIDS. 2010 Jan 28;24(3):427-35. doi: 10.1097/QAD.0b013e328334344e. PMID 19910787
- [Background] Fonquernie F, Lacombe K, Vincensini JP, Boccara F, Clozel S, Ayouch Boda A, Bollens D, Campa P, Pacanowski J, Meynard JL, Meyohas MC, Girard PM. How to improve the quality of a disease management program for HIV-infected patients using a computerized data system. The Saint-Antoine Orchestra program. AIDS Care. 2010 May;22(5):588-96. doi: 10.1080/09540120903280893. PMID 20401768
- [Derived] Tomi AL, Sellam J, Lacombe K, Fellahi S, Sebire M, Rey-Jouvin C, Miquel A, Bastard JP, Maheu E, Haugen IK, Felson DT, Capeau J, Girard PM, Berenbaum F, Meynard JL. Increased prevalence and severity of radiographic hand osteoarthritis in patients with HIV-1 infection associated with metabolic syndrome: data from the cross-sectional METAFIB-OA study. Ann Rheum Dis. 2016 Dec;75(12):2101-2107. doi: 10.1136/annrheumdis-2016-209262. Epub 2016 Mar 31. PMID 27034453